CLINICAL TRIAL: NCT07162480
Title: Phase II Trial of Puxitatug Samrotecan (AZD8205) in Advanced, Recurrent or Metastatic (R/M) Aggressive Adenoid Cystic Carcinoma Subtype I (ACC-I)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0803; NCI-2025-06440 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Adenoid Cystic Carcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- P-Sam (Experimental): Participants will receive P-Sam at 2.4 mg/kg intravenously on D1 of a 21-day treatment cycle
  Interventions: Drug: P-Sam

INTERVENTIONS:
Drug: P-Sam — Given by IV

SUMMARY:
Phase II open label study designed to evaluate the efficacy and safety of P-Sam in patients with aggressive, solid, NOTCH mutant or p63 low (B7-H4 high) R/M ACC-I patients.

DETAILED DESCRIPTION:
Primary Objective:

To assess the objective response rate and safety of P-Sam in patients with R/M ACC-I.

Secondary Objectives:

To estimate the disease control rate (DCR) To estimate the median duration of response (DOR) To estimate the median progression-free survival (PFS) To estimate the PFS rate at 3 and 6 months To estimate the median overall survival (OS) To assess patient's quality of life (QoL) during P-Sam therapy

Tertiary/Exploratory Objectives:

To explore tissue and blood-based biomarkers that may predict response to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years with histology-proven advanced, or R/M ACC.
2. Evidence of locally advanced disease not amenable to curative intent surgery or radiotherapy, or recurrent/metastatic disease
3. ACC-I subtype defined by at least one of the following:

   1. Presence of an activating NOTCH mutation per in-house or any CLIA-certified or commercially available next-generation sequencing assay
   2. Solid histology and clinical course characterized by < 3 years from diagnosis to initial recurrence or progression or de novo metastatic disease with extra-pulmonary metastasis
   3. Negative TP63 tumor expression by IHC (<10% of tumor cells)
4. Measurable disease per RECIST 1.1
5. Performance status ECOG of 0 or 1
6. Patient has provided informed consent.
7. Adequate bone marrow, hepatic, and renal function with the most recent laboratory assessments 8. Contraceptive use by the participant or the participant's partner should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   (a) Male participants: (i) Non-sterilized male participants who are sexually active with a female partner of childbearing potential must use a male condom (plus spermicide, if available) from enrollment throughout the study and for 8 months following the last dose of study drug. It is strongly recommended for the female partner of a male participant to also use a highly effective method of contraception throughout this period, as described in Table 3. In addition, male participants must refrain from sperm donation while on study and for 8 months (5 half-lives plus 6 months) following the last dose of study drug.

   (b) Female participants: (i) Females of childbearing potential must have a negative urine or serum pregnancy test prior to receiving the first dose of study drug. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

(ii) Female participants of childbearing potential who are sexually active with a non-sterilized male partner must agree to use one highly effective method of birth control (defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly, from enrollment throughout the study and for 8 months following the last dose of study drug. It is strongly recommended for the male partner of a female participant to also use male condom (plus spermicide, if available) throughout this period. Cessation of contraception after this point should be discussed with a responsible physician.

9. Patients can be treatment-naïve or have received up to 3 lines of prior systemic therapy in the setting ofR/M disease, however, a maximum of two prior lines of chemotherapy or antibody-drug conjugate (ADC) are allowed. Exceptions include prior B7-H4-targeting ADC or any prior agent with a topoisomerase inhibitor

1 mode of action; those represent exclusion criteria (exclusion criteria #18).

Exclusion Criteria:

1. Treatment with any of the following as detailed below in Table 2:

   Table 2 . Washout period from prior therapies Treatment Washout period Nitrosourea or mitomycin C Within 6 weeks prior to the first dose of study intervention Any investigational agents or study drugs from a previous clinical study Within 5 half-lives or 28 days (whichever is shorter) prior to the first dose of study drug Any other anticancer treatment Within the following time periods prior to the first dose of study intervention: Cytotoxic treatment: 21 days Non-cytotoxic drugs: 21 days or 5 half-lives (whichever is shorter) Biological products including immuno-oncology agents: 28 days Radiotherapy Wide field of radiation (including whole brain radiotherapy) within 4 weeks or limited field radiotherapy (including stereotactic radiotherapy or gamma-knife) for palliation is allowed up to 14 days prior to the first dose of study intervention. Participants who have not recovered from radiotherapy-related toxicity will not be eligible Major surgery (as defined by the Investigator) At least 28 days prior to the first dose of study intervention
2. Unresolved toxicities of Grade ≥ 2 (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE version 5.0) from prior therapy (excluding vitiligo, alopecia, endocrine disorders that are controlled with replacement hormone therapy, and lymphopenia unless it is accompanied by clinical signs of infection or the indication for prophylaxis with antibiotic/antiviral/antifungal therapy). Participants with chemotherapy-induced Grade 2 neuropathy may be eligible at discretion of the Investigator.
3. Active infection, including tuberculosis, SARS-CoV-2, and known infections with hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency. Participants with a past or resolved HBV/HCV infection are eligible if all the following criteria are met:

   1. Negative for HBsAg and positive for total hepatitis B core antibody (anti-HBc) or Positive for HBsAg, but for > 6 months have had normal transaminases and HBV DNA levels between 0-2000 IU/mL (inactive carrier state) and willing to start and maintain antiviral treatment for at least the duration of the study.
   2. HBV DNA levels > 2000 IU/mL but on prophylactic antiviral treatment for the past 3 months and will maintain the antiviral treatment during the study.
   3. Participants testing positive for HCV antibody are eligible only if the polymerase chain reaction test result is negative for HCV RNA.
4. Has a history of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
5. Has clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder or any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement or prior pneumonectomy (complete) or require supplemental oxygen (including intermittent or discretionary use).
6. Patients with history of myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML) or with features suggestive of MDS/AML (as determined by prior diagnostic investigation). Specific screening for MDS/AML is not required.
7. Participants with any of the following cardiac criteria:

   1. History of clinically significant arrhythmia (such as multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (NCI CTCAE version 5.0 Grade 3); symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia.

      NOTE: abnormalities in serum electrolytes that can increase the risk of arrhythmic events (ie, sodium, potassium, calcium, magnesium) should be corrected before starting the study intervention
   2. Uncontrolled hypertension.
   3. Acute coronary syndrome/acute myocardial infarction, unstable angina pectoris, coronary intervention procedure with percutaneous coronary intervention, or coronary artery bypass grafting within 6 months of the start of study treatment.
   4. History of brain perfusion problems (eg, carotid stenosis) or stroke, or transient ischemic attack in the last 6 months prior to screening.
   5. Symptomatic heart failure (as defined by New York Heart Association class ≥ 2).
   6. Prior or current cardiomyopathy.
   7. Severe valvular heart disease.
   8. Resting corrected QT interval using Fridericia's formula (QTcF) > 470 msec
   9. Any factors that increase the risk of corrected QT (interval) (QTc) prolongation or risk of arrhythmic events such as heart failure, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age.
   10. Concomitant medications known to prolong QTc should be used with caution and cannot be used starting with the first dose of study intervention or during the scheduled ECG assessments (see << https://www.crediblemeds.org/ >>).
8. Active CNS disease (patients with asymptomatic or treated CNS lesions who have been off corticosteroids, radiation, or other CNS-directed therapy for at least 4 weeks prior to start of study treatment are not considered active)
9. Uncontrolled intercurrent illness within the last 12 months of start of study treatment, including but not limited to serious chronic GI conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the participant to give written informed consent.
10. Has substance abuse or any other medical conditions that would increase the safety risk to the participant or interfere with participation of the participant or evaluation of the clinical study in the opinion of the Investigator.
11. Receipt of live attenuated vaccine within 30 days prior to the first dose of study intervention. Note:

    Participants, if enrolled, should not receive live attenuated vaccine whilst receiving study intervention and up to 30 days after the last dose of study intervention. Participants can receive COVID-19 vaccines, at the discretion of the Investigator, following a benefit/risk evaluation for the individual participant and in accordance with local rules and regulations and vaccination guidelines.

    Note: If a COVID-19 vaccine is administered it should be done > 72 hours prior to study intervention initiation.
12. For women only - currently pregnant (confirmed with positive pregnancy test), lactating, breastfeeding, or intend to become pregnant during the study.
13. Red blood cell transfusion dependence, defined as requiring more than 2 units of packed RBC transfusions during the 4-week period prior to screening.
14. Current participation in another interventional clinical study
15. History of previous malignancy other than malignancy treated with curative intent and low risk of recurrence. Patients with the following diagnoses represents an exception and may enroll if ≥ 2 years with no evidence of active disease before the first dose of the study drug or if treatment is not indicated:

    1. Non-melanoma skin cancers with no current evidence of disease
    2. Melanoma in situ with no current evidence of disease
    3. Treated or localized, low-risk, cancer of the prostate with prostate-specific antigen of <1 ng/mL
    4. Treated or localized well-differentiated thyroid cancer (stage I)
    5. Cervical carcinoma in situ
    6. Treated ductal/lobular carcinoma in situ of the breast
    7. Treated or localized, low grade, renal cell carcinoma (stage I)
16. Known hypersensitivity to any of the study drugs, the metabolites, or formulation excipient
17. Cognitively impaired patients who are incompetent to consent.
18. Prior exposure to a B7-H4 targeting ADC, or any prior agent with a topoisomerase inhibitor 1 mode of action.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Renata Ferrarotto, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org